CLINICAL TRIAL: NCT00193843
Title: Phase III Trial of Surgery Followed by Conventional RT(5fr/Week)Vs.Concurrent Chemo-Radiotherapy Vs.Accelerated RT(6fr/Week)in High Risk, Loco-Regionally Advanced, Stage III&IVA, Resectable, Squamous Cell Carcinomas of Oralcavity
Brief Title: Oral Cancer Adjuvant Therapy (OCAT) Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH/177/2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2005-12-26 (Estimated); Status verified 2005-09

CONDITIONS: Mouth Neoplasms
Keywords: Oral cancer; Head and neck surgery; Accelerated radiotherapy; Chemo-radiotherapy
MeSH Terms: conditions — Mouth Neoplasms

INTERVENTIONS:
Procedure: Post-operative chemoradiotherapy / accelerated radiotherapy

SUMMARY:
To demonstrate whether addition of Concurrent chemotherapy to post-operative adjuvant radiotherapy OR shortening of duration of post-operative radiotherapy, by administering 6 fractions / week instead of 5 fractions / week improves local-regional control and / or overall survival in high risk, locally advanced, resectable, squamous cell carcinoma of oral cavity.

DETAILED DESCRIPTION:
Locally advanced, stage III and IVA, resectable, squamous cell carcinomas of oral cavity are conventionally treated with surgery, followed by post-operative radiotherapy. Local-regional recurrence remains the most frequent cause of failure of this treatment. The results of conventional therapy are dismal with five-year survival of less than 30% and 60-80% incidence of local-regional failure within 3 years. There are various known histological prognostic factors. The local-regional control and overall survival are extremely poor in high risk patients with these poor prognostic factors. In an attempt to improve the outcome of this high risk group, various alternative treatment policies such as addition of chemotherapy to radiotherapy or altered fractionation schedules have been tried. But till date, there is no alternative treatment modality with acceptable toxicity, available for these patients.

Aims Of Study: To demonstrate whether addition of Concurrent chemotherapy to post-operative adjuvant radiotherapy OR shortening of duration of post-operative radiotherapy, by administering 6 fractions / week instead of 5 fractions / week improves local-regional control and / or overall survival in high risk, locally advanced, resectable, squamous cell carcinoma of oral cavity.

Eligibility criteria: Locally advanced, stage III and IVA, resectable, squamous cell carcinomas of oral cavity with one of the following poor prognostic factors extracapsular nodal extension, involvement of > 2 regional lymph nodes, margin of resection with invasive cancer Extensive soft tissue and / or skin infiltration requiring major reconstructive procedure.

Peri-neural invasion with positive lymph node. Lympho-vascular embolisation with positive lymph node.

Trial Design The eligible patients will be randomly allocated to one of the three arms

1. Arm 1 (Control arm): Surgery followed by conventional radiotherapy
2. Arm 2: Surgery followed by Concurrent chemo-radiotherapy
3. Arm 3: Surgery followed by Accelerated radiotherapy

Surgery: Surgery will be same in all three arms. Wide excision tumour with appropriate nodal dissection and reconstruction utilizing accepted criteria for the region involved will be done.

Radiotherapy: Total dose of radiotherapy will be 56 - 60 Gy. Patients in Arms 1 and 2, five fractions per week for six weeks. Patients in Arm 3, six fractions a week for five weeks.

Chemotherapy: Patients in Arm 2 will get weekly chemotherapy (Inj Cisplatin 30 mg / m2)

Stratification: Patients will be stratified according to following factors Site: Gingivo-buccal complex cancers Vs Tongue and Floor of mouth cancers. T stage. N stage. Extra-capsular spread (Peri-nodal extension) Surgical margin Extensive soft tissue infiltration

End points Primary end point: Local-regional failure. Secondary end point: Overall survival. Other parameters to be assessed are Treatment related toxicity Protocol compliance Overall treatment time Quality of life: assessment by EORTC-QLQ-C30 and EORTC-H&N-35 Sample size: 900 pts (300 pts in each arm). Duration of accrual: 7 years. Duration of follow up: 5 years. With minimum follow up of 2 years. Analysis: Intent to treat analysis will be done. Interim analysis will be done after 450 patients (150 pts in each arm)

ELIGIBILITY:
Inclusion Criteria:

Previously untreated, resectable, loco-regionally advanced, stage III & IV, biopsy-proven squamous cell carcinoma of the oral cavity. (Clinically lower stage patients will also be included if upstaged to pathological stage III or IV after Surgery)

One or more of the following must be present:

extracapsular nodal extension, involvement of > 2 regional lymph nodes, margin of resection with invasive cancer (on histopathology) Extensive soft tissue and / or skin infiltration requiring major reconstructive procedure.

Peri-neural invasion with positive lymph node(s). Lymphovascular embolisation with positive lymph node(s). Age > 18. Karnofsky performance status of > 60. WBC > 3500, platelets > 100,000 Serum creatinine < 1.2 mg / m2 Signed study-specific informed consent form. Protocol treatment must begin within 8 weeks surgery.

Exclusion Criteria:

Gross (visible or palpable) residual disease left after surgery. Prior chemotherapy or radiation therapy to the head and neck region.

Evidence of distant metastasis. Any post-operative complication which will delay starting of adjuvant treatment for more than 8 weeks.

Presence of synchronous or concurrent head and neck primary tumors. Prior malignancy within the previous 5 years. Patients who because of their medical status are not candidates for the proposed treatment.

KPS < 60. Age > 65 years. Poor expected follow up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2005-06; Study Completion 2017-06

PRIMARY OUTCOMES:
Local-regional failure

SECONDARY OUTCOMES:
Overall survival
Treatment related toxicity
Protocol compliance
Overall treatment time
Quality of life: assessment by EORTC-QLQ-C30 and EORTC-H&N-35

CONTACTS AND LOCATIONS:
Overall Officials: Mandar S Deshpande, MBBS,MS,DNB, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai 12, Maharashtra, India; Mandar S Deshpande, MBBS,MS,DNB, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai 12 .Maharshtra, India
Locations (1):
- Dr. Mandar. S. Deshpande, Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Laskar SG, Chaukar D, Deshpande M, Chatterjee A, Sinha S, Chakraborty S, Agarwal JP, Gupta T, Budrukkar A, Murthy V, Pai P, Chaturvedi P, Pantvaidya G, Deshmukh A, Nair D, Nair S, Prabhash K, Swain M, Kumar A, Noronha V, Patil V, Joshi A, DCruz A. Oral cavity adjuvant therapy (OCAT) -a phase III, randomized controlled trial of surgery followed by conventional RT (5 fr/wk) versus concurrent CT-RT versus accelerated RT (6fr/wk) in locally advanced, resectable, squamous cell carcinoma of oral cavity. Eur J Cancer. 2023 Mar;181:179-187. doi: 10.1016/j.ejca.2022.12.016. Epub 2022 Dec 26. PMID 36669426